CLINICAL TRIAL: NCT05599594
Title: Effect of Neroli and Lemongrass Oils With Premenstrual Symptoms and Effect on Quality of Life: Randomized Controlled Research
Brief Title: Premenstrual Symptoms and Aromatherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Karataysid
Record Dates: First submitted 2022-04-26; First posted 2022-10-31 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2022-12

CONDITIONS: Premenstrual Syndrome; Aromatherapy
Keywords: Aromatherapy; Premenstrual symptom; Quality of life
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: 3 groups will be formed from the students identified with the symptoms of premenstrual syndrome. 1.Gruba Neroli, 2.Gruba Lemongrass, to Group 3
  (Placebo Group) will be given water vapor and the states of premenstrual syndrome among the groups and the status of premenstrual symptoms will be evaluated. Pre-process pre-test will be applied to all groups. After each application will be tested again. The final test will be applied to each participant's first day of menstruation.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the study, the evaluation and statistical analysis will be blinded. Statistical analyzes will be carried out by a faculty member other than researchers. A non-aware of the experiment and control groups will be aware of the assessment of initiatives. Data entries will be entered with "A", "B" and "C" code without the test or control group specified. Writing the analysis and research report of the data will be carried out to be coded as "A", "B" and "C" group. After the statistical analysis is made and the research report is written, the encoders for the experiment and the control group will be explained by the encoder by the encoder. The data collection tool described below before the venture and the control group will be applied below
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neroli oil (Experimental): Neroli oil improves the quality of life by reducing premenstrual symptoms with relaxing and calming effect.
  Interventions: Other: Aromatherapy
- Lemongrass oil (Experimental): Lemongrass oil improves the quality of life by reducing premenstrual symptoms with relaxing and calming effect.
  Interventions: Other: Aromatherapy

INTERVENTIONS:
Other: Aromatherapy — 6 drops of aromatic oils used by the researcher will be dripped by the aromatic oils to take the fragrance by inhalation for 30 minutes.

SUMMARY:
Aromatherapy is the science of using high concentrated essential oils or essences with distilled high concentration of plants to take advantage of therapeutic properties '' . Essential oils or essences are obtained from various parts of plants (root, leaf, flower, shell, fruit) and therapeutically used for physical and psychological favors. The aromatherapine is a noninvasive process and the convenience of use allows the widespread use of aromatherapy. Aromatic oils can be applied in four basic ways. These are topical (tap, compressed or bath), internal (mouthwash, vaginal or anal wick), mouth (with capsules or honey, alcohol or diluent) and inhalation (inhalation directly or indirectly, steam or vapor ) is the way . Volatile oils that can be applied in various means can reach the neocortex part of the brain directly with the links to the hypothalamus from the limbic system. As a result of the impact of aromatic oils on the central nervous system, relief, sedation or stimulating effects are formed and the energy blockage in the body is broken, due to the information stream reaching the brain with the warning of the central nervous system and the resulting energy is exposed. The improvement process is supported by its exposed energy stream in a balanced way of the relevant organs, and the state of physical and spiritual goodness is emerged. Aromatherapy is also used in the field of women's health as well as many health areas.

DETAILED DESCRIPTION:
Premenstrual syndrome is a health problem characterized by mitigation of symptoms in several days after the beginning of menstruals, or after the beginning of menstruals, which occurs in the Luteal phase of menstrual cycle in the luteal phase . About 80-95% of women complained of premenstrual syndrome complaints. This ratio is affected by physical, cognitive, emotional and behavioral symptoms in different occupational groups in serious dimension, it can negatively affect life from business life to family life, and when it is considered to be repeated each month, the quality of life is negatively affected. In this reason the premenstrual symptoms The minimization of complaints and minimizing complaints constitutes a state of need.

In the studies involved in the literature, women complaining about Premenstrual Syndrome complaints were applied to various essential oils (Rose, Sardinia, Sage, Lavender) aromatherapy and stated that depression, anxiety, anxiety, irritability pain perception decreased by both psychological and physical positive effects.

In Turkey, the trend of traditional and complementary medicine is increasing day by day. However, aromatherapy practices are common in Turkey as well as aromatherapy practices in the world. The aromatic oils are diluted and ready to use are a method in pharmacies, as well as in pharmacies, as well as people want to use and use. The cost of ready-to-use aromatic oils will provide the treatment option to women in the light of new evidence in line with the fact that it is cheap and easily accessible to the study .

ELIGIBILITY:
Inclusion Criteria:

* Premenstrual is at least 5 of the complaints living (self-notice),
* Non-respiratory disease such as asthma, bronchitis (self-notice),
* Not allergic to fat to be used (self-notice),
* Pregnancy or pregnancy doubt (self-notice),
* Diabetes, hypertension without a systemic discomfort (self-notice)

Exclusion Criteria:

* Premenstrual has not experienced complaints,
* Using cigarettes or alcohol,
* With chronic discomfort (respiratory diseases),
* Pregnancy suspected or conceived,
* With a systemic discomfort such as diabetes, hypertension,
* Individuals who do not want to participate in the study

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | 1 year
  A questionnaire with 12 questions was created by the researchers. The filling time of the participants is 5-6 minutes.
Premenstrual Syndrome Scale | 1 year
  Participants in the study will be asked to fill in this scale in the pre-test. Women with premenstrual syndrome will be included in the study.The application of the premenstrual syndrome scale is made by evaluating the person retrospectively, taking into account the "being in the period one week before the period". The total score is obtained from the sum of the scores from all sub-dimensions. A minimum of 44 and a maximum of 220 points can be obtained from the scale. An increase in the score obtained from the scale indicates an increase in the intensity of the symptoms. If the total scale score (220) exceeds 50% (110) in the PMS scale, PMS is considered as "present".

SECONDARY OUTCOMES:
Scale for Coping With Premenstrual Symptoms | 1 year
  Participants will be asked to fill in this scale both in the pretest and the posttest.No evaluation is made on the total score of the Scale for Coping with Premenstrual Symptoms. As the score obtained from the sub-dimensions of the scale increases, coping with premenstrual symptoms increases. The scale structure consisting of thirty-two items explains 38.9% of the variance. In addition, the sub-dimensions of the scale are in a significant relationship with each other, and the correlation coefficients range from 0.188 to 0.518. Cronbach's alpha safety coefficients of the sub-dimensions of the Turkish version of PSSS were ''harm avoidance-0.88'', ''awareness and acceptance of premenstrual changes -0.89'', ''adapting energy -0.75'', ''self-care-0.83''. ' is 'communication-0.86''.
SF-36 Quality of Life Scale | 1 year
  Participants will be asked to fill in this scale both in the pretest and the posttest.The scale consists of eight sub-dimensions for physical function, physical role limitations, emotional role limitations, vitality (life energy), social function, pain, mental health and general perception of health. A separate score is obtained for each subscale. SF-36 evaluates the positive as well as the negative aspects of the health condition. Sub-dimension scores range from 0 to 100. Scores are positively oriented. Increasing score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Füsun SUNAR, Associate Professor, Principal Investigator — Kto Karatay Üniversitesi
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No